CLINICAL TRIAL: NCT05698095
Title: A Phase 1, First-in-human, Double-blind, Placebo-controlled, Randomized, Single- and Multiple-ascending-dose Study to Determine the Safety, Tolerability, and Pharmacokinetics of 5-methoxy-N,N-dimethyltryptamine (5-MeO-DMT) Administered by Intramuscular Injection in Healthy Subjects
Brief Title: Pharmacokinetics, Safety, and Tolerability of Intramuscular 5-MeO-DMT in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: MEO101
Record Dates: First submitted 2023-01-05; First posted 2023-01-26 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pharmacokinetics; Safety; Tolerability
Keywords: 5-MeO-DMT; Psychedelics; Safety; Pharmacokinetics; First-in-human; 5-methoxy-N,N-dimethyltryptamine
MeSH Terms: interventions — Methoxydimethyltryptamines; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study will include separate single- and multiple-dose parts.
  Single-dose part:
  A double-blind, placebo-controlled, randomized, sequential-group design with 5-MeO-DMT administered by intramuscular injection in 6 cohorts of 6 subjects (randomized as 5 active and 1 placebo subject(s) per group).
  Multiple-dose part:
  A double-blind, placebo-controlled, randomized, sequential-group design with 5-MeO-DMT administered by intramuscular injection in up to two doses within a single day (3-hour interval) with two different dose levels (6 subjects per group).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 - 0.5 mg single-dose (Experimental): A single 0.5 mg 5-MeO-DMT or placebo dose administered intramuscularly (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo
- Cohort 2 - 2.5 mg single-dose (Experimental): A single 2.5 mg 5-MeO-DMT or placebo dose administered intramuscularly (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo
- Cohort 3 - 4.5 mg single-dose (Experimental): A single 4.5 mg 5-MeO-DMT or placebo dose administered intramuscularly (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo
- Cohort 4 - 7 mg single-dose (Experimental): A single 7 mg 5-MeO-DMT or placebo dose administered intramuscularly (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo
- Cohort 5 - 10 mg single-dose (Experimental): A single 10 mg 5-MeO-DMT or placebo dose administered intramuscularly (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo
- Cohort 6 - 13 mg single-dose (Experimental): A single 5-MeO-DMT 13 mg or placebo dose administered intramuscularly (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo
- Cohort 7 - multiple-dose, 3 hour interval (Experimental): Administration of up to two 5-MeO-DMT (2.5 mg followed by 4.5 mg) or placebo doses administered intramuscularly within a single day with a 3 hour dose interval (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo
- Cohort 8 - multiple-dose, 3 hour interval (Experimental): Administration of up to two 5-MeO-DMT (2.5 mg followed by 7 mg) or placebo doses administered intramuscularly within a single day with a 3 hour dose interval (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo
- Cohort 9 - multiple-dose, 3 hour interval (Experimental): Administration of up to two 5-MeO-DMT (2.5 mg followed by 10.5 mg) or placebo doses administered intramuscularly within a single day with a 3 hour dose interval (randomized as 5 active and 1 placebo subject).
  Interventions: Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt; Drug: Placebo

INTERVENTIONS:
Drug: 5-methoxy-N,N-dimethyltryptamine succinate salt — The 5-MeO-DMT drug product is comprised of the appropriate concentration of 5-MeO-DMT succinate salt drug substance in solution with 0.9% sodium chloride injection solution (USP) in a 5 mL glass vial, and is administered intramuscularly.
  Other Names: 5-MeO-DMT succinate salt; 5-MeO-DMT
Drug: Placebo — The placebo is commercially available 0.9% sodium chloride solution (USP) for injection. The placebo is provided by the pharmacy in single-use sterile syringes of the appropriate dose.
  Other Names: 0.9% sodium chloride solution (USP)

SUMMARY:
The primary objective of the study is to assess the pharmacokinetics, safety, and tolerability of a single-dose and multiple-doses of 5-MeO-DMT administered by intramuscular (IM) injections in healthy subjects.

DETAILED DESCRIPTION:
This study is a phase 1, first-in-human, double-blind, placebo-controlled, randomized, single-dose and multiple-ascending-dose study of 5-MeO-DMT administered by intramuscular injection in 54 healthy subjects (adult male and/or females, 18-65 years of age). Subjects will be randomized 6:1 to receive 5-MeO-DMT or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female.
* Aged at least 18 years but not older than 65 years, inclusive.
* Body mass index (BMI) within 18.0 kg/m2 to 32.0 kg/m2, inclusive.

Exclusion Criteria:

* History of significant hypersensitivity to the IP or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, or endocrine disorders, as determined by the investigator (or designee).
* Participants who, in the opinion of the investigator (or designee), should not participate in this study.
* Participant is participating in another study with a medical device or IP within the last 30 days prior to first study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events as coded by MedDRA and assessed by CTCAE v4.0 | Up to 30 Days
  Number of participants with TEAEs following administration of 5-MeO-DMT.

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters of 5-MeO-DMT and bufotenine following a single-dose and multiple-doses of 5-MeO-DMT | Up to 24 hours
  For PK analysis, blood samples will be collected before and up to 24 hours after the intramuscular administration of 5-MeO-DMT to determine 5-MeO-DMT and bufotenine serum concentrations.
Urine pharmacokinetic parameters of 5-MeO-DMT and bufotenine following a single-dose and multiple-doses of 5-MeO-DMT | Up to 24 hours
  For PK analysis, urine samples will be collected before and up to 24 hours after the intramuscular administration of 5-MeO-DMT to determine 5-MeO-DMT and bufotenine urine concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Kansas, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reckweg J, Mason NL, van Leeuwen C, Toennes SW, Terwey TH, Ramaekers JG. A Phase 1, Dose-Ranging Study to Assess Safety and Psychoactive Effects of a Vaporized 5-Methoxy-N, N-Dimethyltryptamine Formulation (GH001) in Healthy Volunteers. Front Pharmacol. 2021 Nov 25;12:760671. doi: 10.3389/fphar.2021.760671. eCollection 2021. PMID 34912222
- [Background] Shen HW, Jiang XL, Winter JC, Yu AM. Psychedelic 5-methoxy-N,N-dimethyltryptamine: metabolism, pharmacokinetics, drug interactions, and pharmacological actions. Curr Drug Metab. 2010 Oct;11(8):659-66. doi: 10.2174/138920010794233495. PMID 20942780
- [Background] Barsuglia J, Davis AK, Palmer R, Lancelotta R, Windham-Herman AM, Peterson K, Polanco M, Grant R, Griffiths RR. Intensity of Mystical Experiences Occasioned by 5-MeO-DMT and Comparison With a Prior Psilocybin Study. Front Psychol. 2018 Dec 6;9:2459. doi: 10.3389/fpsyg.2018.02459. eCollection 2018. PMID 30574112
- [Background] Davis AK, Barsuglia JP, Lancelotta R, Grant RM, Renn E. The epidemiology of 5-methoxy- N, N-dimethyltryptamine (5-MeO-DMT) use: Benefits, consequences, patterns of use, subjective effects, and reasons for consumption. J Psychopharmacol. 2018 Jul;32(7):779-792. doi: 10.1177/0269881118769063. Epub 2018 Apr 30. PMID 29708042
- [Background] Ermakova AO, Dunbar F, Rucker J, Johnson MW. A narrative synthesis of research with 5-MeO-DMT. J Psychopharmacol. 2022 Mar;36(3):273-294. doi: 10.1177/02698811211050543. Epub 2021 Oct 19. PMID 34666554
- [Background] Uthaug MV, Lancelotta R, van Oorsouw K, Kuypers KPC, Mason N, Rak J, Sulakova A, Jurok R, Maryska M, Kuchar M, Palenicek T, Riba J, Ramaekers JG. A single inhalation of vapor from dried toad secretion containing 5-methoxy-N,N-dimethyltryptamine (5-MeO-DMT) in a naturalistic setting is related to sustained enhancement of satisfaction with life, mindfulness-related capacities, and a decrement of psychopathological symptoms. Psychopharmacology (Berl). 2019 Sep;236(9):2653-2666. doi: 10.1007/s00213-019-05236-w. Epub 2019 Apr 13. PMID 30982127
- [Background] Sherwood AM, Claveau R, Lancelotta R, Kaylo KW, Lenoch K. Synthesis and Characterization of 5-MeO-DMT Succinate for Clinical Use. ACS Omega. 2020 Dec 2;5(49):32067-32075. doi: 10.1021/acsomega.0c05099. eCollection 2020 Dec 15. PMID 33344861